CLINICAL TRIAL: NCT02779959
Title: Buccal Prochlorperazine Versus Intravenous Prochlorperazine for Migraine Headaches, a RCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, David Tanen, Professor of Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30590-01
Record Dates: First submitted 2016-05-17; First posted 2016-05-23 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Prochlorperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buccal Prochlorperazine (Experimental): Experimental arm of two buccally absorbable prochlorperazine tablets (6 mg) plus 2 cc IV saline
  Interventions: Drug: Prochlorperazine
- Intravenous Prochlorperazine (Active Comparator): Accepted Standard of care receiving 10 mg (2 cc) of intravenous prochlorperazine plus two saccharin absorbable placebo tablets.
  Interventions: Drug: Prochlorperazine

INTERVENTIONS:
Drug: Prochlorperazine

SUMMARY:
Headache is a common presenting complaint to the emergency department accounting for 1-2% of patient visits. Of these headaches, approximately 90% are migraine, tension headache, or combined presentations. The most commonly used migraine therapy in the ED is intravenous prochlorperazine, but its administration requires close nursing observation, a bed, and the insertion of an intravenous catheter. Buccal prochlorperazine represents an alternative form of delivery that enables rapid achievement of therapeutic blood levels and may lead to symptom resolution. In a randomized, controlled, prospective study,the investigators plan to assess the efficacy of buccal versus intravenous prochlorperazine for the initial emergency department treatment of migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-65 years of age evaluated in the emergency department at Harbor-UCLA with migraine headache as defined by the Headache Classification Committee of the International Headache Society. (Patients must have had at least one prior similar headache, with or without nausea, vomiting, aura, photophobia, or phonophobia).
* Only subjects able to consent to treatment will be included.

Exclusion Criteria:

Patients with the following conditions:

* pregnancy
* breastfeeding
* fever greater or equal to 100.4 degrees
* diastolic blood pressure of 105 or higher
* altered mental status
* meningeal signs
* suspicion for intracranial process requiring further investigation
* known allergy to prochlorperazine
* the use of ergotamines, antiemetics, antipsychotics or sedatives in the previous 24 hours of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in median pian VAS score | From Time 0 (baseline) to Time 60 minutes after administration of medication
  Primary end point will be a detectable difference in the median pain VAS score recorded from Time 0 (baseline) to Time 60 minutes (conclusion of the study) for each of the two groups.

SECONDARY OUTCOMES:
Change in median sedation VAS scores | From Time 0 (baseline) to Time 60 minutes after administration of medication
  Secondary endpoints will include a detectable difference in median sedation VAS scale from Time 0 (baseline) to Time 60 minutes (conclusion of the study for each of the two groups.
Change in median nausea VAS scores | From Time 0 (baseline) to Time 60 minutes after administration of medication
  Secondary endpoints will include a detectable difference in median nausea VAS scale from Time 0 (baseline) to Time 60 minutes (conclusion of the study for each of the two groups.
Rescue Medication | At the conclusion of the study (60 minutes)
  Comparison between groups for the need for rescue medication as determined by the primary care provider.
Follow-up for persistence or recurrence of headache | 24 -48 hours
  Using a Pain Relief Scale, subjects will be contacted by telephone at 24 - 48 hours after the conclusion of the study and asked to rate their current headache pain.

CONTACTS AND LOCATIONS:
Overall Officials: David Tanen, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No